CLINICAL TRIAL: NCT00767845
Title: PROSTATE CANCER SYMPTOM MANAGEMENT FOR LOW LITERACY MEN
Brief Title: Symptom Management in African-American Men With Localized Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were enrolled here or at UCSF.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Latini, Assistant Professor, Baylor College of Medicine
Other Study IDs: CDR0000600455; BCM-H-19323
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire/survey administration

SUMMARY:
RATIONALE: Gathering information about symptom management from patients with localized prostate cancer may help doctors improve patients' quality of life.

PURPOSE: This clinical trial is studying symptom management in African-American men with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop a symptom management intervention for African-American men treated for localized prostate cancer, with a particular emphasis on low health literacy men.

OUTLINE: Participants are interviewed by the principal investigator over the phone or meet the principal investigator at the Veterans Administration prostate cancer clinic. If the interview is conducted in the clinic, it is held in a private room in the clinic.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven localized prostate cancer

  * Has received treatment for prostate cancer
* Patient self-identifies as being of African-American descent

PATIENT CHARACTERISTICS:

* Able to speak and read in English
* Has an address in order to receive study materials by mail (a street address or post office box)
* Has either a telephone in order to be interviewed OR is able to meet the principal investigator at the Veterans Administration prostate clinic and be interviewed there

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Symptom management taxonomy

CONTACTS AND LOCATIONS:
Overall Officials: David M. Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas, United States